CLINICAL TRIAL: NCT03113383
Title: Visceral Manifold Study for the Repair of Thoracoabdominal Aortic Aneurysms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device recalled by the manufacturer
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Thomas Naslund, Professor Vascular Surgery, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161627
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Results first posted 2022-02-10 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Thoracoabdominal Aortic Aneurysm
Keywords: Thoracoabdominal Aortic Aneurysm; Endovascular Aneurysm Repair; Stent-Graft
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Primary Arm (Experimental): Use of the thoracic bifurcation and the visceral manifold to repair thoracoabdominal aortic aneurysms in patients having appropriate anatomy.
  Interventions: Device: Thoracoabdominal Aortic Aneurysm Repair
- Expanded Selection Arm (Experimental): Use of the thoracic bifurcation and the visceral manifold to repair thoracoabdominal aortic aneurysms in patients having appropriate anatomy.
  Interventions: Device: Thoracoabdominal Aortic Aneurysm Repair

INTERVENTIONS:
Device: Thoracoabdominal Aortic Aneurysm Repair — Thoracoabdominal aortic aneurysm repair

SUMMARY:
The primary objective of the clinical investigation is to assess the use of the the Visceral Manifold Thoracoabdominal Aortic Aneurysms (VTAAA) stent graft system to repair thoracoabdominal aortic aneurysms in patients having appropriate anatomy. The primary intent of the study is to assess safety (i.e. freedom from major adverse events (MAE) at 30 days) and preliminary effectiveness (i.e., treatment success and technical success) of the device (i.e., the proportion of treatment group subjects that achieve and maintain treatment success at one year).

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the safety of this device as there are no or very limited devices and clinical options available for this patient population. The primary safety endpoint of this study is safety freedom from major adverse events (MAE) at 30 days or during hospitalization if this exceeds 30 days. Major adverse events include death, bowel ischemia, myocardial infarction, paraplegia, renal failure, respiratory failure, and stroke. The primary safety endpoint will be analyzed to determine statistical significance when compared to a target performance goal. A literature review of outcomes of open surgical repair was used to create the performance goal as there is not a comparable endovascular option to use for analysis. The performance goal was selected based on the range of subjects experiencing a major adverse event at 30 days. The range was calculated based on assumptions of the minimum and maximum number of subjects experiencing at least one MAE in the historical open surgical repair group . Based on the literature reviewed and the above assumptions the range of subjects experiencing at least one MAE in the open surgical repair group is 30.5% to 77.4%.

The primary effectiveness endpoint is the proportion of the study subjects with treatment success at 1 year. The data will be presented as quality outcomes with the number of study subjects with treatment success compared to the overall patient population.

Additionally, data outcomes from this study will be entered into a common vascular database so that data can be pooled with other PS-IDEs. This would provide consistent reporting across the PS-IDEs. Additionally, the PS-IDEs will be evaluating the same device and endpoints to allow for a pool-ability of data across the sites.

The pooled data will be separated into two separate study arms: primary study arm and expanded selection arm.

ELIGIBILITY:
Primary Arm

General Inclusion Criteria:

* A patient may be entered into the study if the patient has at least one of the following:

  * An aneurysm with a maximum diameter of greater than or equal to 5.5 cm or 2 times the normal diameter just proximal to the aneurysm using orthogonal (i.e., perpendicular to the centerline) measurements
  * Aneurysm with a history of growth greater than or equal to 0.5 cm in 6 months
  * Saccular aneurysm deemed at significant risk for rupture
  * Symptomatic aneurysm greater than 4.5 cm
* Axillary or brachial and iliac or femoral access vessel morphology that is compatible with vascular access techniques, devices or accessories, with or without use of a surgical conduit
* Proximal landing zone for the thoracic bifurcation stent graft that has:

  * Greater than or equal to 2.5 cm of nonaneurysmal aortic segment including previously placed graft material (neck) distal to the left subclavian artery (LSA) diameter in the range of 26-42 mm
  * Adequate distance from the celiac artery, in order to accommodate cannulation from the antegrade access point when considering the total deployed length of the thoracic bifurcation and visceral manifold
  * Minimum branch vessel diameter greater than 5 mm
* Iliac artery or aortic distal fixation site, including both native tissue and previously placed graft, greater than or equal to 15 mm in length and diameter in the range of 8 - 25 mm
* Age: greater than or equal to 18 years old
* Life expectancy: greater than 1 year

Exclusion Criteria:

* Patient is a good candidate for and elects for open surgical repair
* Can be treated in accordance with the instructions for use with a legally marketed endovascular device
* Is eligible for enrollment in a manufacturer-sponsored IDE at the investigational site
* Unwilling to comply with the follow-up schedule
* Inability or refusal to give informed consent
* Urgent or emergent presentation
* Patient is pregnant or breastfeeding
* Patient has a contained rupture
* Patient has a ruptured aneurysm
* Patient has a dissection in the portion of the aorta intended to be treated
* Obstructive stenting of any or all of the visceral vessels
* Poor performance status including two major system failures (including but not limited to cardiovascular, pulmonary, renal, hepatobiliary, and neuromuscular)

Medical Exclusion Criteria

* Known sensitivities or allergies to the materials of construction of the devices, including nitinol (Nickel: Titanium) polyester, platinum-iridium, polytetrafluoroethylene (PTFE), platinum, gold, polyethylene, or stainless steel.
* Known hypersensitivity or contraindication to anticoagulation or contrast media that cannot be adequately medically managed
* Uncorrectable coagulopathy
* Body habitus that would inhibit x-ray visualization of the aorta or exceeds the safe capacity of the equipment
* Patient has had a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned less than 30 days of the endovascular repair
* Unstable angina (defined as angina with a progressive increase in symptoms, new onset at rest or nocturnal angina)
* Systemic or local infection that may increase the risk of endovascular graft infection
* Baseline creatinine greater than or equal to 2.0 mg/dL
* History of connective tissue disorders (e.g., Marfan Syndrome in the primary arm only, not applicable for patients in the the expanded access arm, Ehler's Danlos Syndrome)
* Prior aneurysm repair that would involve relining of the previously placed graft material requiring placement of the investigational system in a landing zone that expands beyond any limits of the previously placed graft material

Anatomical exclusion criteria:

* Minimum branch vessel diameter less than 5 mm
* Thrombus or excessive calcification in the proximal aortic neck
* Anatomy that would not allow maintenance of at least one patent hypogastric artery
* Anatomy that would not allow primary or assisted patency of the left subclavian artery

Expanded Selection Arm Inclusion Criteria

* Patient that meets the criteria for inclusion in the primary study arm but has one or more of the following criteria which would exclude them from the primary study arm:
* Minimum branch vessel diameters <less than 5mm
* Urgent or emergent presentation
* Patient has a contained rupture
* Patient has a ruptured aneurysm
* Patient has a type B dissection (subacute or chronic) in the portion of the aorta intended to be treated
* Poor performance status including two major system failures (including but not limited to cardiovascular, pulmonary, renal, hepatobiliary, and neuromuscular)
* Baseline creatinine greater than greater than or equal to 2.0 mg/dL
* Anatomy that does not allow for maintenance of at least one hypogastric artery
* Anatomy that does not allow primary or assisted patency of the left subclavian artery
* Prior aneurysm repair that would involve relining of the previously placed graft material requiring placement of the investigational system in a landing zone that expands beyond any limits of the previously placed graft material
* Obstructive stenting of any or all of the visceral vessels

Or

* A patient that meets the criteria for inclusion into the primary study arm and:
* Would not be eligible for the primary study arm per a documented reason other than those outlined above, and
* Per the opinion of the Principal Investigator, with concurrence of the IRB, alternatives therapies are unsatisfactory and the probable risk of using the investigational device is no greater than the probable risk from the disease or condition.

These will be determined by standard of care assessments of their disease/aneurysm morphology by the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2021-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Naslund, MD, Principal Investigator — Chief, Division of Vascular Surgery
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Data outcomes from this study will be entered into a common vascular database so that data can be pooled with other PS-IDEs. This would provide consistent reporting across the PS-IDEs. Additionally, the PS-IDEs will be evaluating the same device and endpoints to allow for a pool-ability of data across the sites.
  The pooled data will be separated into two separate study arms: primary study arm and expanded selection arm.
Supporting Information: CSR
Time Frame: Upon completion of the study
Access Criteria: Pooled data will be shared with other investigators evaluating the same device and endpoints.

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Primary Arm; Experimental: Expanded Selection Arm: Use of the thoracic bifurcation and the visceral manifold to repair thoracoabdominal aortic aneurysms in patients having appropriate anatomy.
Period: Overall Study
Arm/Group | Experimental: Primary Arm | Experimental: Expanded Selection Arm
Started | 4 | 0
Completed | 0 | 0
Not Completed | 4 | 0
Not completed — Death | 4 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Primary Arm
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint: Freedom From Major Adverse Events
Description: Freedom from major adverse events (MAE) at 30 days.
Time Frame: 30 days
Population: No data was collected.
Arm/Group | Primary Arm | Expanded Selection Arm
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Preliminary Effectiveness
Description: Proportion of subjects treated with the device that achieve and maintain treatment success at 1 year.
Time Frame: 1 year
Population: Data was not collected.
Arm/Group | Primary Arm | Expanded Selection Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Secondary Safety Endpoint:Freedom From Major Adverse Events
Description: Freedom from major adverse events (MAE) at 6 Months.
Time Frame: 6 months
Population: No data collected.
Arm/Group | Primary Arm | Expanded Selection Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Secondary Safety Endpoint: Freedom From Major Adverse Events
Description: Freedom from major adverse events (MAE) at 1 year.
Time Frame: 1 year.
Population: No data collected
Arm/Group | Primary Arm | Expanded Selection Arm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Secondary Safety Endpoint: Freedom From Major Adverse Events
Description: Freedom from major adverse events (MAE) at 2 years.
Time Frame: 2 years.
Population: No data collected
Arm/Group | Primary Arm | Expanded Selection Arm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Secondary Safety Endpoint: Freedom From Major Adverse Events
Description: Freedom from major adverse events (MAE) at 3 years.
Time Frame: 3 years.
Population: No data collected
Arm/Group | Primary Arm | Expanded Selection Arm
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Secondary Safety Endpoint: Freedom From Major Adverse Events
Description: Freedom from major adverse events (MAE) at 4 years.
Time Frame: 4 years.
Population: No data collected
Arm/Group | Primary Arm | Expanded Selection Arm
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Secondary Safety Endpoint: Freedom From Major Adverse Events
Description: Freedom from major adverse events (MAE) at 5 years.
Time Frame: 5 years.
Population: Data were not collected at this time point as the study was terminated before 5 years
Arm/Group | Primary Arm | Expanded Selection Arm
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Secondary Effectiveness Assessment
Description: Proportion of subjects treated with the device that achieve and maintain treatment success at 30 days as defined by aneurysm exclusion.
Time Frame: 30 days.
Population: No participants enrolled in the Expanded Selection Arm
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Arm | Expanded Selection Arm
Number analyzed (Participants) | 4 | 0
Participants | 3 | 0

10. Secondary Outcome: Secondary Effectiveness Assessment
Description: Proportion of subjects treated with the device that achieve and maintain treatment success at 6 months as defined by aneurysm exclusion.
Time Frame: 6 months.
Population: There were no patients alive at 6 months. No data was collected.
Arm/Group | Primary Arm | Expanded Selection Arm
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Secondary Effectiveness Assessment
Description: Proportion of subjects treated with the device that achieve and maintain treatment success at 2 years as defined by aneurysm exclusion.
Time Frame: 2 years.
Population: There were no patients alive at 2 years. No data was collected.
Arm/Group | Primary Arm | Expanded Selection Arm
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Secondary Effectiveness Assessment
Description: Proportion of subjects treated with the device that achieve and maintain treatment success at 3 years as defined by aneurysm exclusion.
Time Frame: 3 years.
Population: There were no patients alive at 3 years. No data was collected.
Arm/Group | Primary Arm | Expanded Selection Arm
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Secondary Effectiveness Assessment
Description: Proportion of subjects treated with the device that achieve and maintain treatment success at 4 years as define by aneurysm exclusion.
Time Frame: 4 years.
Population: There were no patients alive at 4 years. No data was collected.
Arm/Group | Primary Arm | Expanded Selection Arm
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Secondary Effectiveness Assessment
Description: Proportion of subjects treated with the device that achieve and maintain treatment success at 5 years as define by aneurysm exclusion.
Time Frame: 5 years.
Population: There were no patients alive at 5 years. No data was collected.
Arm/Group | Primary Arm | Expanded Selection Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 Years and 2 months
Description: Adverse events were assessed from enrollment until 30 days after procedure. All-Cause Mortality was from date of procedure up to 4 years and 2 months
Arm/Group | Experimental: Primary Arm | Experimental: Expanded Selection Arm
All-Cause Mortality (participants affected / at risk) | 4/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/4 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Primary Arm (N=4) | Experimental: Expanded Selection Arm (N=0)
Multi-organ failure - (General disorders) | 2 (2) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT03113383/Prot_SAP_000.pdf